CLINICAL TRIAL: NCT01656213
Title: Randomised Control Trial for Improving Functional Outcome From Stroke in End Stage Renal Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12/LO/0087
Record Dates: First submitted 2012-07-11; First posted 2012-08-02 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2012-07

CONDITIONS: Stroke; End Stage Renal Disease
Keywords: Stroke; End Stage Renal Disease; Recovery; Haemodialysis
MeSH Terms: conditions — Stroke; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- visual-feedback handgrip exercise (Experimental): Subjects allocated to treatment will be trained in the laptop-based exercise that takes 20 minutes/session. Subjects will be encouraged to perform the exercise 2-3 times per dialysis session
  Interventions: Device: Computer-based target pursuit task (created using E-Prime software) and visual-feedback handgrip force transducer (CurrentDesigns 2012).
- Control Arm (No Intervention): 60 similar ESRD stroke patients will be randomly assigned to the non-intervention arm. These patients will receive standard advice during dialysis (rest or gentle activity, e.g. reading).
  Note that both groups of patients will also receive standard multidisciplinary rehabilitation care following a stroke, including therapy sessions at times other than receiving dialysis

INTERVENTIONS:
Device: Computer-based target pursuit task (created using E-Prime software) and visual-feedback handgrip force transducer (CurrentDesigns 2012). — Subjects will be encouraged to perform the exercise 2-3 times per dialysis session depending upon mood, although will be permitted to skip sessions if they do not feel well or motivated. The laptop program time-stamps each session, and records a time-series of duration, force and accuracy of hand grip.
  Arms: visual-feedback handgrip exercise

SUMMARY:
TITLE Randomised Control Trial (RCT) for improving functional outcome from stroke in renal disease patients DESIGN Eandomised Conrol Study AIMS

1. Undertake detailed characterisation of stroke (including recently developed imaging techniques at Imperial) of stroke in renal disease patients including clinical, imaging and epidemiological data
2. To Investigate if passive intervention using hand grip device during dialysis sessions will improve functional outcome from stroke in end stage renal disease patients.

OUTCOME MEASURES

1. Primary outcome:. 3 months change in Upper-Extremity Fugl-Meyer scores.
2. Secondary outcome: 3 months change in NIHS & Bartel scores

POPULATION Ischaemic and haemorrhagic stroke patients with renal disease treated at Hammersmith's Hospital's renal Unit. .

ELIGIBILITY Data of all patients with renal disease and imaging proven stroke will be retrospectively analysed. RCT will be conducted on End Stage Renal Disease patients with acute (<7 days) stroke affecting arm.

DURATION 2 years

DETAILED DESCRIPTION:
Randomised Control Trial. ESRD patients on dialysis who have suffered an acute (<7 days) stroke (ischaemic/haemorrhagic) and predicted to have the worst likely outcome (see above) will be recruited for this RCT. Stroke patients will be randomly assigned to the intervention (60 patients) or standard treatment (60 patients) arms (power calculation below). Patients will have detailed demographic information documented. In addition, type, frequency and length of time on dialysis will be noted. Pre-/post- Upper-Extremity Fugl-Meyer scores will be undertaken (sensitive measure of arm motor function).

60 patients will be randomly allocated to the visual-feedback handgrip (affected arm) exercise that we have developed in-house (using Current Designs hand-grip force transducer, and E-Prime software). Subjects allocated to treatment will be trained in the laptop-based exercise that takes 20 minutes/session. Subjects will be encouraged to perform the exercise 2-3 times per dialysis session depending upon mood, although will be permitted to skip sessions if they do not feel well or motivated. The laptop program time-stamps each session, and records a time-series of duration, force and accuracy of hand grip.

Non-intervention. 60 similar ESRD stroke patients will be randomly assigned to the non-intervention arm. These patients will receive standard advice during dialysis (rest or gentle activity, e.g. reading).

Note that both groups of patients will also receive standard multidisciplinary rehabilitation care following a stroke, including therapy sessions at times other than receiving dialysis

3.1 STUDY OUTCOME MEASURES Primary outcome. 3 months change in Upper-Extremity Fugl-Meyer scores. Secondary outcome: 3 months changes in NIHS & Bartel scores

* PARTICIPANT ENTRY

4.1 PRE-REGISTRATION EVALUATIONS We will recruit patients, who suffered from imaging proven, acute stroke affecting arm, while undergoing maintenance haemodialysis at the Imperial College NHS Trust as well as retrospectively analyse data of all patients with renal disease and stroke treated at Hammersmith Hospital

4.2 INCLUSION CRITERIA Patients with imaging proven, acute (<7days) stroke affecting arm, on maintenance dialysis will be recruited into the RCT. Patients have to be able to consent for the study either in writing, verbally or nonverbally in presence of a witness. We will retrospectively analyse the database of all renal disease patients with stroke. This data was collected by Hammersmith Hospital's Renal Team. In case of non-English speaking patients we will use Hospital's interpreter's services to explain the study to the patient, obtain their consent and train them in using the device. .

4.3 EXCLUSION CRITERIA Patients unwilling to give consent, patients unable to use hand grip tool due to severe hand weakness (MRC 0/5), patients unable to understand English or their native language due to receptive aphasia, dementia. Patients with arteriovenous fistula in the affected arm will be excluded from the trial

4.4 WITHDRAWAL CRITERIA Patients unwilling to further participate in the study. Patients, who lose capacity to consent during the study. Patient experiencing side effects. In these cases the data collected will be used for final analysis but no new data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with imaging proven, acute (<7days) stroke affecting arm, on maintenance dialysis will be recruited into the RCT. Patients have to be able to consent for the study either in writing, verbally or nonverbally in presence of a witness. We will retrospectively analyse the database of all renal disease patients with stroke. This data was collected by Hammersmith Hospital's Renal Team. In case of non-English speaking patients we will use Hospital's interpreter's services to explain the study to the patient, obtain their consent and train them in using the device

Exclusion Criteria:

* Patients unwilling to give consent, patients unable to use hand grip tool due to severe hand weakness (MRC 0/5), patients unable to understand English or their native language due to receptive aphasia, dementia. Patients with arteriovenous fistula in the affected arm will be excluded from the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Upper-Extremity Fugl-Meyer scores | 3 months
  sensitive measure of arm motor function

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz pucek, M.D., Principal Investigator — Imperial College London
Locations (1):
- Imperial College NHS Trust, London, London, United Kingdom